CLINICAL TRIAL: NCT06243250
Title: Integrated Precision Imaging for Immune-related Adverse Events: Hyperpolarized 13C-MRI and Metabolomics
Brief Title: Hyperpolarized 13C-MRI and Metabolomics for Immune-related Adverse Events
Acronym: DNP_irAE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: DNP_irAE
Record Dates: First submitted 2024-01-17; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Immune-related Adverse Event
Keywords: Immune Checkpoint inhibitor; Immune-related Adverse Event; Spleen; Hyperpolarized 13C-MRI; Pyruvate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- with irAE: Cancer patients who develop irAE after ICIs treatment.
  Interventions: Diagnostic Test: Hyperpolarized 13C-MRI
- without irAE: Cancer patients who do not develop irAE after 3 months of ICIs treatment.
  Interventions: Diagnostic Test: Hyperpolarized 13C-MRI
- healthy volunteer: Healthy volunteer.
  Interventions: Diagnostic Test: Hyperpolarized 13C-MRI

INTERVENTIONS:
Diagnostic Test: Hyperpolarized 13C-MRI — Metabolic MRI using IV injection of hyperpolarized [1-13C]pyruvate.

SUMMARY:
This project investigates immune-related adverse events (irAEs) in cancer patients treated with immune checkpoint inhibitors (ICIs), focusing on metabolic changes. It explores how glucose metabolism in the spleen, which mirrors immune activity, might predict irAEs. Using advanced imaging like hyperpolarized (HP) 13C-MRI and metabolomics, the study aims to detect metabolic flux in the spleen, potentially offering early prediction and risk categorization of irAEs. The 3-year study will involve 30 cancer patients on ICIs, comparing those with and without irAEs. It hypothesizes that splenic metabolic alterations seen in HP 13C-MRI can forecast and categorize irAE severity, improving our understanding of irAEs and potentially guiding new treatments.

DETAILED DESCRIPTION:
Immune-related adverse events (irAEs) have become clinical challenges with the exponential increase in the use of immune checkpoint inhibitors (ICIs) in medical oncology. irAEs can be fulminant and fatal, requiring personalized management. Early prediction and accurate risk categorization of irAEs are urgently needed to tailor patient management. Glucose metabolism in the spleen may reflect immune activity and has been used to predict tumor response to ICIs. Since the underlying mechanism of irAEs is similar to ICIs tumor response, the splenic metabolism is a potential biomarker for irAEs.

This project is novel because it aims to investigate irAEs from the perspective of metabolism by integrating hyperpolarized (HP) 13C-MRI, metabolomics, and MR fingerprinting (MRF). HP 13C-MRI is a new non-invasive, real-time dynamic imaging technique used to detect the metabolic flux in vivo. Dynamic nuclear polarization (DNP) is a hyperpolarization technique that increases the signal of 13C-labeled probes by up to 50,000-fold. With DNP, [1-13C]pyruvate can be used to probe various metabolic pathways, including its conversion to lactate (anaerobic glycolysis), alanine (transamination), and bicarbonate (indirect marker for TCA cycle). These specific metabolic alterations have been used to characterize the functions of immune cells; thus, they may also reflect the splenic immune activity in patients with irAEs. Additionally, NMR-based metabolomics analyses of patients' serum and urine will provide a more global view of metabolic changes of whole human body. Furthermore, the observed metabolic alterations can be translated into multiparametric tissue properties obtained by MRF.

The investigator design a 3-year project with a non-randomized, two group assignment observational study design. This research will include 30 cancer patients receiving ICIs. Twenty patients experiencing acute phase irAEs (grade 2 or higher) and 10 patients not experiencing irAEs after 14 weeks of treatment will be recruited for this prospective single institutional study. A dedicated multidiscipline immune-oncologic board will screen patients who develop irAEs, which include colitis, endocrinopathy, hepatitis, pneumonitis, and skin toxicity. The diagnosis of the irAEs is determined by clinical history, laboratory values, standard-of-care imaging, and histopathologic features when biopsy is necessary. Participants eligible for this study will undergo investigative exams including HP 13C-MRI, metabolomics, and MRF.

The investigator hypothesize that the spleen immune activity interrogated using HP 13C-MRI can predict the occurrence of irAEs. Additionally, the level of splenic metabolic alterations based on HP 13C-MRI will be correlated to the clinical severity of irAEs, providing additional risk categorization for irAEs. Moreover, by establishing metabolic information and tissue characteristics obtained by MRF, the dynamic changes of immune activity may be monitored by the quantifiable and reproducible tissue properties. Finally, by combining HP 13C-MRI and metabolomics, the investigator will have a better understanding of the pathophysiology of irAEs from the perspective of metabolism, which may lead to the development of new therapy.

ELIGIBILITY:
Inclusion Criteria

Patients undergoing ICIs:

1. Inform consent obtained.
2. Patients more than or equal to 20-year-old.
3. Patients developing IRAEs or not, including but not limited to the following events: colitis、endocrinopathy、hepatitis、pneumonitis、skin toxicity.

Healthy volunteers:

1. Inform consent obtained.
2. Patients more than or equal to 20-year-old.

Exclusion Criteria

Patients undergoing ICIs:

1. Life-threatening irAEs (CTCAE ≥ grade 4).
2. Abnormal spleen attributable to other diseases (e.g., liver cirrhosis related splenomegaly or primary/metastatic splenic tumors).
3. Pregnant or breast-feeding women.
4. Contraindication to MRI study (e.g., claustrophobia or non-removable devices or implants that are incompatible with MRI).
5. Intercurrent illness that will affect the compliance of the patient during the MRI study (e.g., active infection, symptomatic congestive heart failure, uncontrollable angina, arrhythmia, psychiatric disorders, dyspnea, or diarrhea).
6. Severe hepatic dysfunction (alkaline phosphatase/aspartate aminotransferase/alanine aminotransferase >20 × upper limit of normal [ULN] or bilirubin > 10 × ULN).
7. Severe renal impairment (eGFR <30 ml/min/1.73m2).

Healthy volunteers:

1. Pregnant or breast-feeding women.
2. Contraindication to MRI study (e.g., claustrophobia or non-removable devices or implants that are incompatible with MRI).
3. Body mass index (BMI) >35 kg/m2.
4. Significant clinical history of any kind, including but not limited to the following conditions: diabetes mellitus (DM), hypertension (HTN), heart disease, liver disease, kidney disease, blood disorders, immune system-related diseases, etc.
5. Need for medication due to any medical condition within the last 14 days.
6. History of substance abuse (e.g., alcoholism with blood alcohol concentration ≥0.08%).

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A delicate multidiscipline immune-oncologic board will screen the patients who develop acute phase irAEs, which include colitis, endocrinopathy, hepatitis, pneumonitis, and skin toxicity. The diagnosis of the irAEs is determined by clinical, laboratory, standard-of-care imaging, and histopathologic features when biopsy is necessary.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Metabolic activity in spleen measured as pyruvate-to-lactate conversion rate | Data analysis within 7 days after HP 13C-MRI
  The pyruvate-to-lactate conversion calculated by kinetic modeling-based conversion rate of pyruvate-to-lactate (kPL) and model-free metric (signal-to-noise ratio and area-under-curve).

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Chieh Lai, MD, Principal Investigator — Chang Gung Memorial Hospital, Link
Locations (1):
- Chang Gung Memorial hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No